CLINICAL TRIAL: NCT06915428
Title: Personalized Toolkit Building a Comprehensive Approach to Resource Optimization and Empowerment in Pregnancy & Beyond (PTBCARE+) A Randomized Controlled Trial (RCT) of Personalized Care for Prenatal Stress Reduction and Preterm Birth Disparities Prevention
Brief Title: Personalized Care for Prenatal Stress Reduction & Prevention of Preterm Birth (PTB) Disparities
Acronym: PTBCARE+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-1779; R01MD017947 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-04-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth Complication; Preterm Birth; Preterm Birth Recurrence; Preeclampsia; Preeclampsia (PE); Hypertensive Disorders of Pregnancy; Support Program; Stress; Resilience, Psychological; Empowerment, Patient; Emotional Stress; Pregnancy; Pregnancy Complications; Pregnancy Induced Hypertension; Neonates and Preterm Infants; Cervical Insufficiency; Social Determinants of Health (SDOH); Cervical Shortening; Disparities in Pregnancy Complications; Disparities; Prenatal Care; Care Coordination
Keywords: PTBCARE+; pregnancy-related disparities; patient support program; enhanced prenatal care
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia; Patient Participation; Stress, Psychological; Pregnancy Complications; Hypertension, Pregnancy-Induced; Uterine Cervical Incompetence | interventions — myotrophin; Amyloid; Sleep; Meditation; Aspirin

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study. Specifically, after written, informed consent is obtained, each participant will be randomized, in a 2:1 ratio, to receive the Personalized Toolkit Building a Comprehensive Approach to Resource optimization and Empowerment in Pregnancy & Beyond (PTBCARE+) support program vs. usual prenatal care. The randomization sequence will be generated using an adaptive biased coin technique. Participants remain in their assigned group without opportunity for crossover later in the study.
Masking Description: Lab personnel who receive, process, and analyze study samples are blinded to the study group assignments of participants. They will receive samples labeled only with study identification (ID) number and no participant identifiers, ensuring they remain unaware of which participants belong to which study groups. This blinding helps maintain the integrity of the trial by preventing any potential bias in the handling and analysis of the samples or the reporting of the results of biologic assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program (Active Comparator): The UNC Personalized Toolkit Building a Comprehensive Approach to Resource optimization and Empowerment in Pregnancy & Beyond (PTBCARE+) program is a multifaceted, personalized support program designed to help pregnant people at high risk for preterm birth. It enhances the prenatal care experience by adding extensive support resources.
  Interventions: Behavioral: Care coordination; Behavioral: Electronic massage; Behavioral: support gift #1; Behavioral: Support gift #2; Behavioral: Support gift #3; Behavioral: Support gift #4; Behavioral: Additional PTBCARE+ support; Behavioral: Stress reduction toolkit - Visit 1 (V1); Behavioral: PTBCARE+ mobile application (app) and website; Behavioral: Sleep, meditation, and Wellness app; Behavioral: Emergency low blood sugar kit; Behavioral: Low dose aspirin (LDA); Behavioral: Visit #2 Stress Reduction Toolkit
- Usual Prenatal Care (No Intervention): Participants who are randomized to receive usual care will not receive the PTBCARE+ program. Research team members may contact participants only to remind them of study activities, and will conduct standard in-person follow-up visits per study protocol, but will not provide any additional information or support. Usual care participants will receive standardized resources offered to all prenatal patients in clinic per clinical provider discretion.

INTERVENTIONS:
Behavioral: Care coordination — Research team members will serve as research assistants and will also function as perinatal care coordinators.
  In the care coordination role, team members will provide emotional support, liaise with clinical staff, and execute regularly scheduled check-ins with each study participant. Team members also assist with helping participants with logistics, obtaining and remembering to take prescribed medications, and other similar related activities. Participants receive access to contact the research assistant / care coordinator by text, email, phone, or through the electronic medical record participant portal.
  - Per protocol, the research staff will meet in person with participants at least twice (visit 1, visit 2) during pregnancy and once postpartum (0-10 weeks after delivery, for most participants).
  Research staff may also meet in person with participants prior to visit 1 for recruitment/enrollment purposes.
  Other Names: PTBCARE+
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Electronic massage — Participant is given the option to receive a 15-minute electronic massage / relaxation session in clinic via (a) a specialized massage chair or (b) a massage pad that is placed on top of a standard recliner chair.
  * the electronic massages provide gentle massages and are safe for most people to use throughout pregnancy.
  * participants are always be in control of the massage experience and will be given instructions on how to stop the massage at any time.
  * participants are advised to consult the primary obstetric provider before using the massage chair regarding any specific concerns or questions
  * during the session, participants may view relaxation videos (from free, publicly available sites online).
    * participants may choose to sign up for massage(s) at any obstetric visit in the clinic between visit 1 and delivery.
  Other Names: Massage chair; Relaxation session
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: support gift #1 — * Small gift packet with encouraging items (example of items = coloring kit, tea lights, stickers, bookmarks, keychain fidget toy, printed support index cards, and other similar items).
  * Given between 14+0 and 23+6 weeks gestation at time of routine prenatal appointment
  Other Names: cool calm and collected support gift
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Support gift #2 — * Small gift packet with encouraging items (example of items = coloring kit, tea lights, stickers, bookmarks, keychain fidget toy, printed support index cards, and other similar items).
  * Given between 18+0 and 27+6 weeks gestation at time of routine prenatal appointment
  Other Names: Keep moving forward support gift
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Support gift #3 — * Small gift packet with encouraging items (example of items = coloring kit, tea lights, stickers, bookmarks, keychain fidget toy, printed support index cards, and other similar items).
  * Given between 22+0 and 29+6 weeks gestation at time of routine prenatal appointment
  Other Names: Small acts, big impact: pass it on
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Support gift #4 — * Small gift packet with encouraging items (example of items = coloring kit, tea lights, stickers, bookmarks, keychain fidget toy, printed support index cards, and other similar items).
  * Given between 26+0 and 33+6 weeks gestation at time of routine prenatal appointment
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Additional PTBCARE+ support — Additional benefits / support items and support elements are provided to some participants on an "as needed" basis, per study protocol.
  * Information / details intentionally withheld and not made public in order to preserve the scientific validity of the study and protect the rights of the research participants
  * participant eligibility for additional resources as a part of the PTBCARE+ program will be determined by the research staff on the day of Visit 1 after initial set of surveys are completed, and is per protocol
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Stress reduction toolkit - Visit 1 (V1) — In person check-in with research team member re: participant's needs; research team member provides support.
  Physical items that are included as part of this visit include:
  Tote bag with the following stress reduction items or similar:
  * eye mask
  * set of pocket index cards, printed back and front, on a variety of topics that influence pregnancy health, ranging from physical to emotional/mental
  * water bottles
  * small notebook
  * pill minder case
  * magnet and business card for Health Resources and Services Administration (HRSA) national maternal mental health hotline
  * log in codes for electronic resources
  * initial handouts with self care plan, introduction to stress reduction toolkit, etc.
  Other Names: V1 Stress toolkit
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: PTBCARE+ mobile application (app) and website — Comprehensive, study-specific app that is available as a website or as a downloadable application that includes personalized, interactive modules and resources
  * no study related materials are available without a password
  * goal is to collate reputable sources of information to make investigating things online easier
  * includes optional educational modules for participants
  * also includes option of entering stress, well-being, blood sugar, blood pressure, etc. values with option to easily download recorded values for patient's clinical team
  * available online (computer/laptop), tablet, or smart phone. can be downloaded as a progressive web application (PWA) to a local device and used without internet access
  * Electronic access to the PTBCARE+ website will continue through 10 weeks postpartum unless the participant delivered <16+0 weeks gestation in which case access will continue through 4 weeks postpartum
  Other Names: PTBCARE+ website; PTBCARE+ app
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Sleep, meditation, and Wellness app — * complimentary one-year subscription to Aura - an 'all-in-one' wellbeing app that contains an enormous library of meditations, stories, breath work, work wellness, music, sounds, and more!
  * Participants can access this app as needed throughout pregnancy and beyond, for up to one year after the date of enrollment
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Emergency low blood sugar kit — Pouch contains:
  * printed index card with information about signs and symptoms of low blood sugar
  * printed index card with information about what to do if blood sugar is low
  * 2-3 non-perishable, individually wrapped over the counter candy / glucose-raising options; use for low blood sugar treatment is described on the card
  Only participants who have a diagnosis of diabetes mellitus or glucose intolerance AND have been prescribed an oral medication for blood sugar control or have been prescribed insulin are eligible to receive this.
  Each participant can receive a maximum of two kits during pregnancy; first at enrollment, and the other at visit 2 or until delivery
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Low dose aspirin (LDA) — * Bottle of 90-100 pills (depending on manufacturer)
  * Provided at Visit 1 (after randomization)
  * Patients who received a bottle of low-dose aspirin at Visit 1 are offered a 2nd bottle at Visit 2.
  All patients whose provider recommends or prescribes either 81mg or 162mg of LDA during pregnancy are offered LDA as described herein. LDA must be on the patient's med list or specific notes from the patient's prenatal provider must explicitly note that it is recommended the patient take LDA in pregnancy for it to be offered. Individuals who are receiving LDA due to participation in another study are not eligible to receive LDA from PTBCARE+
  Please note that this is listed as a "behavioral" intervention rather than "drug" intervention because the rational behind providing this over the counter medication is to help make the participant's life easier, and the focus is not on the efficacy of LDA. As such, it is being provided as a behavioral intervention.
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program
Behavioral: Visit #2 Stress Reduction Toolkit — In person check-in with research team member re: participant's needs; research team member provides support.
  Physical items that are included as part of this visit include the following stress reduction items or similar:
  1. Frame + ultrasound photo + certificate of achievement!
     * Picture from anatomy ultrasound (or other subsequent ultrasound) is downloaded, printed, and placed in frame.
     * Certificate of achievement is printed and placed on other side of frame with ultrasound photo
  2. other small items including stickers, printed index cards with supportive messaging, etc.
  Other Names: Celebrate Today, Believe in Tomorrow
  Arms: Personalized Toolkit Building a Comprehensive Approach to Resource (PTBCARE+) Support Program

SUMMARY:
The goal of this clinical trial is to learn if a personalized prenatal support program [(Personalized Toolkit Building a Comprehensive Approach to Resource optimization and Empowerment in Pregnancy & Beyond, (PTBCARE+)] works to lower stress and lower the risk of early delivery in pregnant individuals at high-risk for delivering preterm. The main question[s] it aims to answer are:

* Does the PTBCARE+ patient support program lower patient-reported stress levels during pregnancy?
* Does the PTBCARE+ patient support program improve biologic measures of stress during pregnancy?
* Does the PTBCARE+ patient support program result in a higher chance of delivering a healthy baby at or close to full term?

Researchers will compare people who participate in the PTBCARE+ patient support program to those receive usual care to see if the PTBCARE+ patient support program lowers patient-reported stress, improves biologic measures of stress, and increases the chance of delivering a healthy baby at or close to full term.

Participants will be randomly assigned to receive the PTBCARE+ patient support program or usual prenatal care.

All participants will be asked to:

* complete 2 study visits during pregnancy - including completing electronic surveys, providing a blood and urine sample, measuring the heart rate variability by a clip or the ear or finger, and body composition evaluation using a simple scale-like device.
* complete one study visit postpartum that includes completing electronic surveys, and measuring heart rate variability. Blood and urine sample collection and body composition evaluation via InBody scale are optional at the postpartum visit.

People who are randomly assigned to receive the PTBCARE+ support program will receive several resources to help them during pregnancy. These things include items such as:

* a stress reduction toolkit;
* access to an online website that can also be downloaded as a smart phone app;
* the option to receive an electronic massage while in clinic, and more.
* additional support gifts provided at routine clinical appointments

People who are randomly assigned to receive usual prenatal care will not receive any additional support resources from the study during pregnancy.

DETAILED DESCRIPTION:
This project addresses the major public health problem of preterm birth (PTB), delivery <37 weeks, by deploying a novel, personalized, comprehensive 3-tier PTB prevention program [University of North Carolina (UNC) PTBCARE+]. PTB affects 1 in 10 infants born in the United States (US) and is the leading cause of neonatal morbidity and mortality; survivors are at high risk for lifelong adverse health sequelae. Stress is an established risk factor for both spontaneous PTB (sPTB) and medically indicated PTB miPTB). Of significant public health concern, Black patients have 49% higher rates of PTB, are more likely to have early PTB, and increased perceived stress in pregnancy compared to patients of other races. Stress may alter biology, including stress-related gene expression in maternal blood and allostatic load index. Evidence from other fields of medicine supports incorporation of both stress reduction programs and 'patient navigators' as effective approaches to improve health outcomes, and data in obstetrics supports improved outcomes with PTB specialty clinics. However, such programs are not routinely employed in obstetrics. The effect of a specialty prenatal care program targeting stress reduction as a strategy to reduce PTB and PTB disparities remains unknown, representing a critical knowledge gap.

The central hypothesis of this project is that enrollment in a personalized, comprehensive PTB support program (UNC PTBCARE+) is associated with reduced perceived stress, stress-related gene expression, allostatic load, and lower rates of PTB <35 weeks. This hypothesis is supported by published and preliminary data as follows: First, UNC pregnant patients at high risk for PTB have high rates of stress and life stressors (e.g., financial insecurity, racism). Second, biologic stress markers including gene transcript levels differ by PTB status in mid-pregnancy blood. Third, specialty PTB care reduces stress in a NC cohort. Building upon prior work and that of others, this exciting proposal evaluates the efficacy of the novel UNC PTBCARE+ program.

The investigation focus on PTB <35 weeks due to its relative frequency, higher association with neonatal morbidity and mortality as compared to later PTB, to include PTB in the 34th week of gestation (because the delivery gestational age considered 'standard of care' for delivery among individuals with stable but severe preeclampsia and preterm membrane rupture), and to align with multiple other published PTB RCTs. This study will recruit 1,350 pregnant patients between 8+0 and 19+6 weeks gestation with an elevated a priori risk of either medically-indicated preterm birth or spontaneous preterm birth. Subjects will be randomized 2:1 to receive UNC PTBCARE+ vs. usual care. Randomization will be stratified based on maternal race and ethnicity (individuals who identify only as White and non-Hispanic vs. individuals who identify as belonging to one or more other races and/or Hispanic ethnicity and (b) perceived stress scores (those with perceived stress scores ≥20 vs. those with lower perceived stress scores scores).

All participants, regardless of randomization assignment, will have 2 study visits during pregnancy.

* Visit 1 (V1) will occur at randomization, 8+0 - 19+6 weeks gestation.
* Visit 2 (V2) will occur in mid pregnancy, between 22+0 and 29+6 weeks gestation.

At both visits, patients will complete validated surveys evaluating a broad spectrum of stressors, discrimination, adverse childhood experiences, perceived social support, resiliency, medication barriers and adherence, care access and satisfaction,, intervention fidelity and sustainability, use of stress relief modalities, and have blood collected to measure biologic stress markers.

The UNC PTBCARE+ program is personalized. All patients randomized to UNC PTBCARE+ receive a stress reduction toolkit and will work with a PTB Care Coordinator who will provide support, facilitate clinician-prescribed medical care, and serve as a patient-provider liaison. Additional benefits / support items and support elements are provided to some participants on an "as needed" basis, per study protocol, and are not included in the initial registration to preserve scientific integrity and protect the rights of research participants. This study registration will be updated with complete intervention details after the study is fully enrolled and all participants have delivered.

Psychosocial and financial stressor screening results from V1 will determine UNC PTBCARE+ tier assignment. Thus, participants are randomized only after Visit 1 surveys are completed.

This solutions-oriented RCT of UNC PTBCARE+ vs. usual care provides an ideal forum to test the primary hypothesis and study stress-related PTB pathophysiology through the following Aims:

* Aim 1. Evaluate the effects of the UNC PTBCARE+ program on perceived stress and resilience in pregnant patients at high risk for PTB. Hypothesis: Patients randomized to UNC PTBCARE+ will have lower levels of perceived stress and higher levels of resilience at V2 vs. V1; those randomized to usual care will have no change.
* Aim 2. Quantify the extent to which the UNC PTBCARE+ program is associated with improved biologic stress measures during pregnancy. Hypothesis: Patients randomized to UNC PTBCARE+ will have reduced stress-related gene expression and allostatic load scores in maternal blood at V2 vs. V1 compared to those randomized to usual care who will have no change, increasing insight into PTB pathophysiology.
* Aim 3. Determine the effects of the UNC PTBCARE+ program on PTB <35 weeks. Hypothesis: Patients randomized to UNC PTBCARE+ will have lower rates of early PTB compared to those randomized to usual care.

This study provides tangible, personalized solutions to the major public health problem of PTB and carries enormous potential to provide generalizable, low-risk strategies to reduce PTB and related disparities.

ELIGIBILITY:
Inclusion Criteria:

1. Viable, singleton pregnancy, 8+0 to 19+6 weeks, dated by last menstrual period ± ultrasound using standard obstetric criteria per American College of Obstetricians and Gynecologists.

   Gestational age at first ultrasound by last menstrual period (LMP) / Ultrasound method / Measurement agreement with LMP required • Up to 8 weeks 6 days / crown rump length / ± 5 days
   * 9 weeks 0 days to 13 weeks 6 days / crown rump length / ± 7 days
   * 14 weeks 0 days to 15 weeks 6 days / standard fetal biometry / ± 7 days
   * 16 weeks 0 days to 19 weeks 6 days / standard fetal biometry / ± 10 days
   * Gestational dating / fetal viability must be confirmed by ultrasound prior to enrollment / randomization.
   * Ultrasound report must include documentation of normal fetal heart rate of ≥ 120 beats per minute, or subsequent medical record documentation of auscultation of fetal heart rate ≥ 120 beats per minute.
   * Viability must be confirmed / re-confirmed within 7 days of randomization.

   If initial consent occurs early in pregnancy and V1/randomization occur later, viability must be reconfirmed to ensure ongoing eligibility prior to initiating V1 activities (including surveys) and proceeding with randomization.
2. No signs or symptoms of, or clinical diagnosis of, evolving miscarriage, active preterm labor, preterm prelabor rupture of membranes at the time of enrollment.

   * Cervical dilation at the time of enrollment is an exclusion criterion. However, cervical evaluation and digital cervical exam is not required prior to enrollment.

     (3a) High a priori risk for medically indicated preterm birth - must meet at least one of the following 3 criteria (maternal medical history, prior pregnancy history, or moderate risk factor history)
   * miPTB criteria #1: Maternal Medical History - any one of the following:

     o Known chronic hypertension requiring medications in the 3 months prior to conception or prior to 22 weeks gestation.

     o At least 2 blood pressure readings 6 hours apart, <20 weeks gestation, with systolic ≥ 130 mmHg or diastolic ≥ 80 mmHg *regardless of need for medication or formal diagnosis of hypertension in chart*

     o Pre-gestational diabetes mellitus.
     * Diabetes diagnosed <20 weeks gestation.
     * Maternal chronic or sub-acute renal disease, including chronic kidney failure, chronic renal insufficiency, glomerulonephritis, lupus nephritis, defined as any:

       *biopsy proven chronic renal disease history; and/or

       *serum creatinine ≥ 1.1 mg/dL at any time during pregnancy prior to enrollment, in the absence of other identifiable transient factors per clinician's assessment (e.g., extreme dehydration, cystitis, pyelonephritis); and/or

       *chronic proteinuria, defined as baseline urine protein:creatinine ratio ≥ 0.30 mg/dL or 24 hour total urine protein ≥ 300 mg in the absence of other identifiable transient factors per clinician's assessment (e.g., extreme dehydration, cystitis, pyelonephritis)

       *Systemic Lupus Erythematosus
       * Antiphospholipid Antibody Syndrome
   * miPTB criteria #2: Prior pregnancy history - any ONE of the following: o Previous pregnancy complicated by preeclampsia or hypertensive disorders of pregnancy at any gestational age, in a singleton gestation; the fetus must not have had major structural anomalies or aneuploidy.

     o Previous history of stillbirth ≥ 16+0 weeks in a singleton gestation; the fetus must not have had major structural anomalies or aneuploidy. The stillbirth etiology must not have been attributed to physical trauma (e.g., domestic violence, motor vehicle accident) or illicit drug use (e.g., cocaine use leading to abruption and stillbirth).
   * miPTB criteria #3: Any two or more of the following moderate risk factors: o Nulliparity, defined as no prior pregnancy to reach at least 20 weeks gestation note that this is the traditional / classic definition of 'nulliparous' and that there is overlap between nulliparity as defined this way and 'preterm birth' due to cervical insufficiency, which allows for deliveries in the 16-19 week gestational age range to be considered as 'preterm births'

     o Obesity: current or pre-pregnancy body mass index ≥30 kg/m^2

     o Family history: first degree relative with a history of preeclampsia

     o Advanced maternal age: maternal age ≥ 35 years at estimated date of confinement

     o Prior adverse obstetric history - one or more of the following:

     - history of low birth weight or small for gestational age baby in a singleton gestation, defined as weight <10% for gestational age and fetal sex; the fetus must not have had major structural anomalies or aneuploidy.

     - history of adverse pregnancy outcome in a singleton gestation; the fetus must not have had major structural anomalies or aneuploidy.

     o Long interpregnancy interval: ≥ 10 year (3650 day) pregnancy interval, defined as the time (in days) between the date of delivery of the last pregnancy to reach ≥ 20 weeks gestation and the first day of the last menstrual period for the current pregnancy.

     o Black or African-American race (as a proxy for underlying racism) - self-reported. Participants who self-identify as being of more than one racial group will be considered to be of Black race for the purposes of this criterion if one of the racial groups is Black or African-American.
     * Low socioeconomic status, defined as one or more of the following: housing or food insecurity noted in chart within the last year, self-pay or Medicaid insurance, less than high school education

and/or

(3b) High a priori risk for spontaneous preterm birth - must meet at least one of the following 2 criteria (prior pregnancy history or current pregnancy course)

* sPTB criteria #1: Prior pregnancy history

  * EITHER a history of a delivery of a singleton, non-anomalous baby between 16+0 and 34+6 weeks gestation or delivery of a twin, non-anomalous pregnancy between 160 /7and 276 /7 weeks gestation due to spontaneous preterm labor, preterm premature rupture of membranes, cervical insufficiency, or placental abruption - Chart documentation of prior preterm birth, the gestational age of the prior preterm birth (referred to as the 'qualifying delivery') should be determined. If the gestational age at delivery is obtained directly from the medical record and more than one gestational age appears, the greater of the two will be used assuming that neither is the 'source document' (i.e. an ultrasound report with a due date, a c-section report, a delivery note, etc).

Use the following table as a validation of the previous delivery. For example, if the infant was male and weighed more than 2763 grams (6 pounds, 1.5 ounces) then the patient would be ineligible based on history of a preterm birth criteria. This table should only be used to determine whether the qualifying delivery is most likely to be preterm less than 35 weeks gestation when the gestational age CANNOT be verified/calculated by review of the medical records or is not available in the medical records.

Gestational age 90th percentile - boys 90th percentile - girls 33 weeks > 2488g 5 lbs 7.8 oz > 2116g 4 lbs 10.6 oz 34 weeks > 2763g 6 lbs 1.5 oz > 2379g 5 lbs 3.9 oz 35 weeks > 3084g 6 lbs 12.8 oz > 2661g 5 lbs 13.9 oz

* Documented history of a prior pregnancy complicated by asymptomatic cervical shortening <25mm between 16+0 and 23+6 weeks gestation or cervical dilation ≥ 0.5cm requiring cervical cerclage placement prior to 24+0 weeks gestation, even if delivery ultimately occurred ≥ 35 weeks gestation or at term.

  • sPTB criteria #2: Current pregnancy course
* Asymptomatic cervical shortening <25mm in the current pregnancy, diagnosed by transvaginal ultrasound that is performed ≥14+0 weeks gestation, per Registered Diagnostic Medical Sonographer(RDMS) certified Sonographer or physician with transvaginal ultrasound training program (or similar) qualifications
* Cervical cerclage in situ in the current pregnancy due to concern for risk of preterm birth, at the discretion of the primary obstetric provider

  (4) Ability to provide written, informed consent in English or Spanish

  (5) Planned prenatal care at the University of North Carolina at Chapel Hill obstetrics clinics and planned delivery at the University of North Carolina Women's Hospital (Chapel Hill, NC).

Exclusion Criteria:

1. Participation in another intervention based clinical trial during pregnancy that is deemed, at the discretion of the investigative team for the current study or the other concurrent study, to conflict with this research and/or confound the study results.

   o There are some concurrent studies, even those designed to test an intervention, which may be compatible with the current study; this will be reviewed by the investigative leadership team on a case-by-case basis.
2. Previous participation in the PTBCARE+ program in another pregnancy, with randomization to the PTBCARE+ (active intervention) group.
3. Current, ongoing, illicit drug use ≥ 12 weeks gestation.

   * Use of tobacco and/or marijuana products is not an exclusion.
   * Receiving treatment for opioid use disorder with methadone, suboxone, or similar in an approved treatment program is not an exclusion.
4. History of radical trachelectomy
5. Planned voluntary termination of pregnancy.
6. Heavy vaginal bleeding or large subchorionic hemorrhage - defined as:

   * Bleeding as primary reason for unplanned clinic evaluation or emergency room visit within 14 days of potential enrollment
   * Subjective bleeding accompanied by ≥ 4 point drop in the hematocrit within 14 days of potential enrollment
   * Subchorionic hemorrhage or abruption on formal ultrasound with a volume ≥ 64 cubic cm (4cm x 4cm x 4cm) within 14 days of potential enrollment
7. Major congenital anomaly such as major structural deficit of the heart, lungs, brain, or other major organ system

   1. Mild renal abnormalities, clubfoot, isolated cleft lip/palate, etc. in the fetus are not a reason for exclusion.
   2. Isolated 'soft markers' for aneuploidy (such as choroid plexus cysts, echogenic bowel, etc.) are not a reason for exclusion.
   3. If a major congenital anomaly is diagnosed *after* enrollment, the patient will continue to participate in the study, however, the investigators will plan to analyze the study results with and without these individuals included.
8. Positive aneuploidy screening test (traditional biochemical assay, e.g., quad screen - risk of aneuploidy of 1:25 or higher or cell free deoxynucleic acid (DNA) test result that is screen positive for trisomy 13, trisomy 18, trisomy 21, or sex chromosome abnormality) in the absence of definitive fetal karyotype evaluation.

   * Definitive fetal karyotype evaluation can only be obtained through direct testing of the tissue from the conceptus - by chorionic villus sampling or amniocentesis during pregnancy.
   * The term "suspected aneuploidy" is commonly used in the medical record but this is not a diagnosis and by itself is not informative and not an exclusion criteria.
9. Cystic hygroma or abnormally thickened nuchal translucency ≥ 3 mm at any time in the current gestation, regardless of subsequent diagnostic testing results.

   * Note that a cystic hygroma remains an exclusion criterion regardless of subsequent diagnostic testing results because fetuses with this history carry an elevated risk of major congenital heart disease.
   * Fetal echocardiogram is most accurately performed at 22-24 weeks gestation, which is later than the enrollment gestational age window.
10. Polyhydramnios at or prior to enrollment.

    o Polyhydramnios is defined as a maximum vertical pocket ≥ 8.0 cm, given that polyhydramnios <22 weeks has a high likelihood of being associated with congenital anomalies/aneuploidy and/or preterm birth due to preterm prelabor rupture of membranes.
11. For potential participants who meet eligibility criteria ONLY due to prior spontaneous or medically indicated preterm birth: if the prior preterm birth was in a pregnancy complicated by twins, confirmed fetal aneuploidy, or major congenital fetal anomalies in the absence of another pregnancy meeting inclusion criteria they are not eligible.
12. Known HIV positive with viral load greater than 1,000 copies/mL or cluster of differentiation 4 (CD4) count less than 350/mm^3
13. Unwillingness to undergo randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1228 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported Perceived Stress Scores | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Perceived Stress Scale participant survey
  * Scores range 0-40
  * Higher scores = higher stress
Self-reported resilience scores | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Brief Resilience Scale validated participant survey
  * score range = 1-5
  * higher scores = higher resilience
Maternal blood-based stress-related gene transcript levels | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Each participant's fold change in blood-based stress-related gene transcript levels during pregnancy, calculated as a ratio: (visit 2 gene expression - visit 1 gene expression) divided by visit 1 gene expression.
Number of participants with preterm birth or fetal death at 14 weeks 0 days or greater and less than 35 weeks gestation | Between 14 weeks 0 days and 35 weeks 0 days gestation (delivery at 34 weeks 6 days gestation meets the primary outcome; delivery at 35 weeks 0 days gestation does not) , a period of up to 27 weeks from enrollment.
  Number of participants who either delivered or experienced a fetal death at a gestational age between 14 weeks 0 days and 35 weeks 0 days gestation. Pregnancies that are lost in the first trimester (prior to 14 weeks of gestation) are excluded from analysis.

SECONDARY OUTCOMES:
Self-reported (subjective) allostatic load | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Allostatic load = balance between stress and stress-protective factors. This is a single outcome determined by a comprehensive, study-specific calculation from weighted normalized (0-1 scale) data from participant surveys.
  Subjective allostatic load = [(Normalized Stress - Normalized Stress-protective factors)/2]
  * score range -1 to +1
  * higher scores = higher allostatic load (more stress than protective factors)
Self-reported composite "negative" stress | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Subjectively reported composite "negative" stress, which is a single outcome measure calculated by considering participant responses on three surveys. Each survey score total is normalized on a 0-1 scale based on each individual's score in relation to the max possible score for that survey. The 3 normalized scores are then averaged to obtain the single composite negative stress score (range is 0-1), whereby a higher scores = higher negative stress.
Number of participants with composite severe maternal morbidity | Enrollment through the postpartum followup period of 10 weeks after delivery, a period of up to 45 weeks from enrollment (assuming latest possible delivery gestational age is 43 weeks)
  Diagnosis of severe maternal morbidity during pregnancy or the initial postpartum period, defined using indicators by the Centers of Disease Control and Prevention (CDC). Individuals who are diagnosed with one or more of the following by a clinician and with appropriate radiologic / laboratory findings to support the diagnosis are considered to have this outcome:
  acute myocardial infarction, aneurysm, acute renal failure, adult respiratory distress syndrome, amniotic fluid embolism, cardiac arrest / ventricular fibrillation, conversion of cardiac rhythm, disseminated intravascular coagulation, eclampsia, heart failure / arrest during surgery or procedure, puerperal cerebrovascular disorders, pulmonary edema / acute heart failure, severe anesthesia complications, sepsis, shock, sickle cell disease with crisis, air and thrombotic embolism, hysterectomy, temporary tracheostomy, or ventilation. Need for blood transfusion is considered separately, as per prior work.
Perceived Social Support scores | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Social support is quantified by the Medical Outcomes Study (MOS) social support survey
  * score range: 0 to 100
  * High score: Indicates a strong perception of social support, with readily available people to provide assistance and emotional support.
  * Low score: Suggests a perceived lack of social support, potentially indicating a need for additional social connections or support systems.
Satisfaction with medical care | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Determined by the self-administered Patient Satisfaction Questionnaire - 18 question (PSQ-18) survey, which measures satisfaction with medical care across 7 different domains: (1) General satisfaction (2) Technical quality; (3) Interpersonal manner; (4) Communication; (5) Financial aspects; (6) Time spent with doctor; (7) Accessibility and convenience
  * score range = 18 to 90
  * score interpretation: a higher score indicates greater patient satisfaction with their healthcare provider
Self-reported anxiety symptoms | Mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Each participant's subjectively reported anxiety, assessed by the self-administered Generalized Anxiety Disorder - 7 (GAD-7) survey
  Score range: 0 to 21 Score interpretation: higher scores = higher anxiety
Self-reported perinatal depression symptoms | Initial pregnancy intake (administered during routine clinical care during pregnancy, as early as 4 weeks pregnant to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 26 weeks from enrollment
  Depression symptoms are assessed by the Edinburgh Postnatal Depression Scale (EPDS).
  Scoring: range 0-30
  Interpretation: higher scores are associated with higher possibility of depression
Self-reported pregnancy experiences | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  The self-administered pregnancy experiences scale and includes:
  * 10 questions on 'Hassles' with a total hassles score ranging from 0 to 30. Higher Scores: Higher scores on the hassles dimension indicate greater perceived stress and negative experiences during pregnancy.
  * 10 questions on 'uplifts' with a total uplifts score ranging from 0 to 30. Higher scores on the uplifts dimension indicate more positive experiences and emotional upliftment.
  The Composite Measure Score=Total Uplifts Score-Total Hassles Score; Score range = -30 to +30. Interpretation: A positive composite score indicates that the positive experiences (uplifts) outweigh the negative experiences (hassles), suggesting a more positive overall pregnancy experience. Conversely, a negative composite score indicates that hassles outweigh uplifts.
Self-assessed generalized self-efficacy | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  The Generalized Self-Efficacy Scale (GSE) is a 10-item, widely used tool to assess an individual's belief in their ability to handle various challenging situations. Each item is rated on a 4-point scale:
  Total Score: The scores for each item are summed to provide a total score, which ranges from 10 to 40.
  Interpretation: Higher Scores: Indicate a stronger belief in one's ability to cope with difficult situations and achieve goals.
  Lower Scores: Suggest lower confidence in one's ability to manage challenges and may indicate a need for interventions to boost self-efficacy.
Self-assessed overall health | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Each participant's change in their perception of their overall physical health, as assessed by the 10 question Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Survey
  Rating: Each item is rated on a 5-point Likert scale. Responses are summed to create raw scores for physical and mental health. Raw scores are converted to T-scores using standardized tables. T-scores have a mean of 50 and a standard deviation (SD) of 10, based on the general population.
  Interpretation:
  T-Scores at 50 are Representative of the average score of the general population.
  Above 50: Indicates better than average health. Below 50: Indicates worse than average health.
Self-reported coping strategies | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Coping strategies are assessed by the participant reported survey, Coping Strategies Inventory - Short Form (CSI-SF). The CSI-SF has 16 items, 4 per each of 4 sub-scales:
  1. Problem-Focused Engagement
  2. Problem-Focused Disengagement
  3. Emotion-Focused Engagement
  4. Emotion-Focused Disengagement
  Total for each subscale = 4-20.
  * Range for positive coping (adding 2 "engagement" sub-scales) is 8-40
  * Range for negative coping (adding 2 "disengagement" sub-scales) is 8-40. The positive coping score is then divided by the negative coping score to provide a ratio of positive to negative coping, ranging from 0.2 to 5.
  Interpretation: Higher scores on each sub-scale indicate more frequent use of that coping strategy. Thus, a higher positive:negative coping strategy ratio suggests a more adaptive/positive coping style whereas lower ratios suggest less adaptive/more negative coping.
Self-assessed overall well-being | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Overall wellbeing is self-assessed by the Positive Emotion, Engagement, Relationships, Meaning, and Accomplishment (PERMA) Profiler, which measures these 5 key well-being domains. The 5 PERMA domains are averaged to provide an assessment of overall health. The instrument also includes measures for Negative Emotion and Health.
  Scoring Range: each PERMA domain is assessed using three items, rated on a scale from 0 (Never) to 10 (Always). Scores for each domain are averaged to provide a domain score. The overall PERMA score is an average of all scores and ranges from 0-10. Negative Emotion and Health are also assessed using three items each, rated on the same 0 to 10 scale, and averaged.
  Scoring Interpretation: Higher scores indicate higher levels of well-being in the respective domain.
Subjective report of physical activity | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Physical activity is quantified by the Pregnancy Physical Activity Questionnaire Short Form (PPAQ-SF).
  Scoring: The 10 question PPAQ-SF measures physical activity across several domains: (1) Household/Caregiving; (2) Occupational; (3) Sports/Exercise; (4) Transportation; (5) Locomotion. Each activity is categorized by intensity:
  Light activities = 1.5-2.9 metabolic equivalents (METs); moderate activities = 3.0-5.9 METs; vigorous activities = ≥ 6.0 METs.
  Score calculation / range / interpretation: MET hours/week = MET value of activity x hours spent on that activity/week. Higher scores = more active. Theoretically, the minimum score is 0 MET hours/week, indicating no physical activity; there is no strict upper limit, but extremely high scores (>10,000) = uncommon, may indicate over-reporting.
Delivery gestational age | From the time of enrollment (if > 14 weeks 0 days) or 14 weeks 0 days to delivery (may occur as late as 43+0 weeks), a period of up to 35 weeks from enrollment
  Participant's delivery gestational age or gestational age at time they are diagnosed with an in-utero fetal death.
  Delivery gestational age is considered continuously, in weeks and days of gestation. Pregnancies that are lost in the first trimester (prior to 14 weeks of gestation) are excluded from analysis. Therefore the possible range of gestational age entries is 14 weeks 0 days (earliest) through 43 weeks 0 days (generally the latest possible gestational age).
Objective allostatic load index | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Each participant's objective allostatic load index will be calculated using clinical parameters including blood pressure, pulse pressure, and body mass index, etc. based on the published literature.
  Score range = normalized, 0 to 100 scale. Score interpretation = higher allostatic load score = higher allostatic load
Number of participants with preterm birth or fetal death less than 37 weeks gestation | Between 14 weeks 0 days and 37 weeks 0 days gestation (delivery at 36 weeks 6 days gestation meets this outcome; delivery at 37 weeks 0 days gestation does not) , a period of up to 29 weeks from enrollment.
  Number of participants who either delivered or experienced a fetal death at a gestational age between 14 weeks 0 days and 37 weeks 0 days gestation. Pregnancies that are lost in the first trimester (prior to 14 weeks of gestation) are excluded from analysis.
Number of participants with preterm birth or fetal death less than 32 weeks gestation | Between 14 weeks 0 days and 37 weeks 0 days gestation (delivery at 31 weeks 6 days gestation meets this outcome; delivery at 32 weeks 0 days gestation does not) , a period of up to 24 weeks from enrollment.
  Number of participants who either delivered or experienced a fetal death at a gestational age between 14 weeks 0 days and 32 weeks 0 days gestation. Pregnancies that are lost in the first trimester (prior to 14 weeks of gestation) are excluded from analysis.
Number of participants with preterm birth or fetal death less than 28 weeks gestation | Between 14 weeks 0 days and 28 weeks 0 days gestation (delivery at 27 weeks 6 days gestation meets this outcome; delivery at 28 weeks 0 days gestation does not) , a period of up to 20 weeks from enrollment.
  Number of participants who either delivered or experienced a fetal death at a gestational age between 14 weeks 0 days and 28 weeks 0 days gestation. Pregnancies that are lost in the first trimester (prior to 14 weeks of gestation) are excluded from analysis.
Number of participants with preterm birth or fetal death less than 24 weeks gestation | Between 14 weeks 0 days and 24 weeks 0 days gestation (delivery at 23 weeks 6 days gestation meets this outcome; delivery at 24 weeks 0 days gestation does not) , a period of up to 16 weeks from enrollment.
  Number of participants who either delivered or experienced a fetal death at a gestational age between 14 weeks 0 days and 24 weeks 0 days gestation. Pregnancies that are lost in the first trimester (prior to 14 weeks of gestation) are excluded from analysis.
Number of participants with composite placental complications | Baseline (Visit 1 - 8+0 to 19+6 weeks) until delivery (may occur as late as 43+0 weeks), a period of up to 35 weeks from enrollment
  Development of placental complications during pregnancy, defined as one or more of the following:
  1. placental abruption (diagnosed clinically) ± birthweight <3% for fetal sex and delivery gestational age ±
  2. diagnosis of hypertensive disorders of pregnancy (including gestational hypertension, chronic hypertension with superimposed preeclampsia, preeclampsia, eclampsia) ±
  3. intrauterine fetal demise
Parasympathetic Nervous System Index | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Parasympathetic Nervous System (PNS) function is assessed using participant heart rate variability data collected using a continuous heart rate sensor (finger or ear clip) using publicly available Kubios heart rate variability software.
  PNS Index range: -5 to +5.
  Interpretation: A PNS index value of zero indicates that the parameters reflecting parasympathetic activity are, on average, equivalent to those of the normal population. Positive index values signify higher parasympathetic nervous system activity and lower stress; lower values indicate lower parasympathetic activity and increased stress.
Sympathetic Nervous System Index | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Sympathetic Nervous System function is assessed via the Sympathetic Nervous System (SNS) Index using participant heart rate variability data collected using a continuous heart rate sensor (finger or ear clip) using publicly available Kubios heart rate variability software.
  SNS Index range: typically -5 to +5, may fall outside of range.
  Interpretation: A SNS index of zero indicates average sympathetic activity compared to the norm. Positive values reflect sympathetic activity levels above the norm, while negative values indicate lower than average activity. During stress or intense exercise, the SNS index can range significantly higher, potentially reaching values between 5 and 35.
Number of participants with composite neonatal morbidity | Neonatal outcomes are evaluated until initial hospital discharge or 45 weeks post menstrual age, a period of up to 37 weeks from maternal enrollment and up to 23 weeks of age for the neonate (if born at 22 weeks 0 days).
  Neonates born to participants are considered to have composite major neonatal morbidity, if, prior to initial hospital discharge from the delivery hospitalization, they are diagnosed by a clinician with one or more of the following diagnoses:
  1. bronchopulmonary dysplasia
  2. intraventricular hemorrhage grade III or IV
  3. periventricular leukomalacia
  4. necrotizing enterocolitis requiring surgery
  5. death
Heart Rate Variability | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Heart Rate Variability (HRV) is assessed using data collected from participants by a continuous heart rate sensor (finger or ear clip) and calculated using publicly available HeartMath / EmWave Pro heart rate variability software.
  HRV values are reported as a continuous integer and range from 1 - 120 (typical expected upper limit, but may be higher in isolated situations).
  Interpretation: Higher HRV: Generally associated with better cardiovascular health and greater resilience to stress.
  Lower HRV: Can indicate higher stress levels, poor cardiovascular health, or other health issues
Number of participants who are diagnosed with hypertensive disorders of pregnancy | Baseline (Visit 1 - 8+0 to 19+6 weeks) until delivery (may occur as late as 43+0 weeks), a period of up to 35 weeks from enrollment
  Development of hypertensive disorders of pregnancy, one of the elements of the composite placental complications (outcome #24), defined as a diagnosis of gestational hypertension, chronic hypertension with superimposed preeclampsia, preeclampsia, and/or eclampsia through the postpartum followup period.

OTHER OUTCOMES:
Level of engagement with PTBCARE+ intervention | Baseline (Visit 1 - 8+0 to 19+6 weeks) until delivery (may occur as late as 43+0 weeks), a period of up to 35 weeks from enrollment
  Considering only those randomized to the PTBCARE+ intervention, the investigators will evaluate the percentage of eligible activities completed considered as a continuous variable (range = 0-100, with higher numbers indicating higher participation and engagement).
Autonomic function evaluation | Baseline (Visit 1 - 8+0 to 19+6 weeks) and mid-pregnancy followup (Visit 2 - 22+0 to 29+6 week), a period of up to 22 weeks from enrollment
  Autonomic function will be calculated by dividing Sympathetic Nervous System (SNS) function index (outcome #26) by Parasympathetic Nervous System (PNS) function index (outcome #27). Values are obtained using participant heart rate variability data collected using a continuous heart rate sensor (finger or ear clip) using publicly available Kubios heart rate variability software.
  This ratio is a continuous variable that will vary based on SNS index value (expected -5 to +5) and PNS index values (expected -5 to +5), and thus will range -25 to +25. Higher values = higher sympathetic nervous system activity (stressed) relative to parasympathetic activity (relaxed).
Interval between study enrollment and delivery or in-utero fetal death. | From the time of enrollment to delivery (may occur as late as 43+0 weeks), a period of up to 35 weeks from enrollment
  The interval between study enrollment and delivery or diagnosis of in utero fetal demise (the period of "latency") will be considered as a continuous variable (in days/weeks), determined by the following formula:
  Participant delivery gestational age or gestational age at time they are diagnosed with an in-utero fetal death minus the gestational age at study enrollment.
  The possible range of values is 0 days (if delivery occurs same day as study enrollment, albeit unlikely) to 35 weeks (245 days) if the participant enrolls at the earliest possible gestational age of 8 weeks 0 days and delivers at 43 weeks 0 days (generally the latest possible gestational age).
Amount of gestational weight gain | Captured at enrollment and at delivery (may occur as late as 43+0 weeks), a period of up to 35 weeks from enrollment
  Amount of weight gained, in pounds, during pregnancy.
  Calculated by considering:
  Last recorded weight during pregnancy minus the pre-pregnancy weight if measured at medical facility / clinic within 3 months' of last menstrual period (LMP) or calculated start of pregnancy using the best estimated date of conception (EDC), or, if this is unavailable, the earliest recorded weight at a medical facility / clinic during pregnancy.
  Considered as a continuous variable, typical expected range -20 pounds to +100 pounds, though outliers may occur. Higher numbers indicate higher weight gain during pregnancy. Negative numbers reflect weight loss during pregnancy.
Level of satisfaction with PTBCARE+ intervention | Enrollment through the postpartum followup period of 10 weeks after delivery, a period of up to 45 weeks from enrollment (assuming latest possible delivery gestational age is 43 weeks)
  Considering only those randomized to the PTBCARE+ intervention, the investigators will evaluate overall participant satisfaction with the intervention using a study-specific survey. Satisfaction scores will be summed and normalized on a scale of 0-100, with higher scores indicating higher satisfaction with the packaged intervention.
Number of participants requiring a blood transfusion during pregnancy or the immediate postpartum time period | Enrollment through the postpartum followup period of 10 weeks after delivery, a period of up to 45 weeks from enrollment (assuming latest possible delivery gestational age is 43 weeks)
  Need for blood transfusion is one of 21 indicators used to identify severe maternal morbidity, as per the Centers of Disease Control and Prevention. However, receiving a blood transfusion can sometimes not accurately reflect a true severe complication on its own. Small blood transfusions may be administered routinely even without a major adverse event, potentially inflating the rate of severe maternal morbidity if included without further context. Thus, need for blood transfusion during pregnancy or the immediate postpartum time period (through the time of discharge from delivery hospitalization), is evaluated separately.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Manuck, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina School of Medicine - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication of initial results provided the investigator who proposes to use the data:
  1. submits a proposal to the study investigative team regarding the planned use of the data, and:
  2. the data analysis plans fall under the scope of written, informed consent as per the participant consent form;
  3. the proposed analysis does not directly conflict with a pre-specified analysis planned by the primary investigative team at UNC;
  4. (as applicable, based on the request) the proposed individual patient data (IPD) request involves a sufficient number of individuals within individual subgroups such that individual participants cannot be readily identified by review of the IPD.
  5. has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable; and
  6. executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1. De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication of initial results provided the investigator who proposes to use the data in accordance with the guidelines outlined above in the plan description.
  2. The study protocol, statistical analysis plan, and informed consent forms will be shared beginning 3 months following delivery of the final study participant, given the importance that several study details are redacted during the study to preserve study integrity and protect research subjects.
Access Criteria: Who will have access?
  * Researchers & Investigators: Qualified researchers/investigators with legitimate scientific requests.
  * Public: Data may be made available to the public, depending on the ethical considerations and the purpose of data request.
  * Access requests will be reviewed by the investigative team to ensure protection of participant privacy is maintained as per the consent form(s) and IRB.
  What will they be able to access?
  * A subset of the "minimum necessary" de-identified data to fulfill the objectives outlined in the requestor's proposal
  * Access to study protocols, statistical analysis plans, and informed consent documents.
  How will they access it?
  - Researchers must submit a formal data access request, similar to request forms that are required to access data through dbGAP and other similar online data repositories.
  Approved individuals will be able to download de-identified data and supporting documentation from a secure online portal.

REFERENCES:
- [Background] Park S, Marcotte R, Staudenmayer J, Sirard J, VanKim N, Pekow P, Strath S, Freedson P, Chasan-Taber L. Validity of the Pregnancy Physical Activity Questionnaire Short Form (PPAQ-SF). Am J Epidemiol. 2024 Oct 2:kwae382. doi: 10.1093/aje/kwae382. Online ahead of print. PMID 39359005
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Hux VJ, Roberts JM. A potential role for allostatic load in preeclampsia. Matern Child Health J. 2015 Mar;19(3):591-7. doi: 10.1007/s10995-014-1543-7. PMID 24939173
- [Background] Heshmati S, Kibrislioglu Uysal N, Kim SH, Oravecz Z, Donaldson SI. Momentary PERMA: An Adapted Measurement Tool for Studying Well-Being in Daily Life. J Happiness Stud. 2023;24(8):2441-2472. doi: 10.1007/s10902-023-00684-w. Epub 2023 Sep 22. PMID 38130904
- [Background] Addison C, Jenkins B, White M. User Manual for Coping Strategies Inventory Short Form (CSI-SF)-The Jackson Heart Study. Int J Environ Res Public Health. 2024 Apr 4;21(4):443. doi: 10.3390/ijerph21040443. PMID 38673353
- [Background] Luszczynska A, Scholz U, Schwarzer R. The general self-efficacy scale: multicultural validation studies. J Psychol. 2005 Sep;139(5):439-57. doi: 10.3200/JRLP.139.5.439-457. PMID 16285214
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Moser A, Stuck AE, Silliman RA, Ganz PA, Clough-Gorr KM. The eight-item modified Medical Outcomes Study Social Support Survey: psychometric evaluation showed excellent performance. J Clin Epidemiol. 2012 Oct;65(10):1107-16. doi: 10.1016/j.jclinepi.2012.04.007. Epub 2012 Jul 20. PMID 22818947
- [Background] Mustillo S, Krieger N, Gunderson EP, Sidney S, McCreath H, Kiefe CI. Self-reported experiences of racial discrimination and Black-White differences in preterm and low-birthweight deliveries: the CARDIA Study. Am J Public Health. 2004 Dec;94(12):2125-31. doi: 10.2105/ajph.94.12.2125. PMID 15569964
- [Background] Hall LA, Williams CA, Greenberg RS. Supports, stressors, and depressive symptoms in low-income mothers of young children. Am J Public Health. 1985 May;75(5):518-22. doi: 10.2105/ajph.75.5.518. PMID 3985241
- [Background] DeFranco EA, Hall ES, Muglia LJ. Racial disparity in previable birth. Am J Obstet Gynecol. 2016 Mar;214(3):394.e1-7. doi: 10.1016/j.ajog.2015.12.034. Epub 2015 Dec 22. PMID 26721776
- [Background] Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep. 2015 Dec;64(12):1-64. PMID 26727629
- [Background] Vianna P, Bauer ME, Dornfeld D, Chies JA. Distress conditions during pregnancy may lead to pre-eclampsia by increasing cortisol levels and altering lymphocyte sensitivity to glucocorticoids. Med Hypotheses. 2011 Aug;77(2):188-91. doi: 10.1016/j.mehy.2011.04.007. Epub 2011 May 6. PMID 21550175
- [Background] Wadhwa PD, Entringer S, Buss C, Lu MC. The contribution of maternal stress to preterm birth: issues and considerations. Clin Perinatol. 2011 Sep;38(3):351-84. doi: 10.1016/j.clp.2011.06.007. PMID 21890014
- [Background] Vohr B. Long-term outcomes of moderately preterm, late preterm, and early term infants. Clin Perinatol. 2013 Dec;40(4):739-51. doi: 10.1016/j.clp.2013.07.006. Epub 2013 Sep 20. PMID 24182959
- [Background] Bodeau-Livinec F, Marlow N, Ancel PY, Kurinczuk JJ, Costeloe K, Kaminski M. Impact of intensive care practices on short-term and long-term outcomes for extremely preterm infants: comparison between the British Isles and France. Pediatrics. 2008 Nov;122(5):e1014-21. doi: 10.1542/peds.2007-2976. PMID 18977951
- [Background] Manuck TA, Sheng X, Yoder BA, Varner MW. Correlation between initial neonatal and early childhood outcomes following preterm birth. Am J Obstet Gynecol. 2014 May;210(5):426.e1-9. doi: 10.1016/j.ajog.2014.01.046. PMID 24793722
- [Background] Manuck TA, Rice MM, Bailit JL, Grobman WA, Reddy UM, Wapner RJ, Thorp JM, Caritis SN, Prasad M, Tita AT, Saade GR, Sorokin Y, Rouse DJ, Blackwell SC, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Preterm neonatal morbidity and mortality by gestational age: a contemporary cohort. Am J Obstet Gynecol. 2016 Jul;215(1):103.e1-103.e14. doi: 10.1016/j.ajog.2016.01.004. Epub 2016 Jan 7. PMID 26772790
- [Background] Russell RB, Green NS, Steiner CA, Meikle S, Howse JL, Poschman K, Dias T, Potetz L, Davidoff MJ, Damus K, Petrini JR. Cost of hospitalization for preterm and low birth weight infants in the United States. Pediatrics. 2007 Jul;120(1):e1-9. doi: 10.1542/peds.2006-2386. PMID 17606536
- See also: Contains study brochure, provided to potentially interested participants — https://www.ptbcare.com/study-brochure
- See also: Health-related social determinants of health including financial stress, as per the NC Department of Health and Human Services consensus — https://www.ncdhhs.gov/about/department-initiatives/healthy-opportunities/screening-questions
- See also: information regarding heart rate variability and health and regarding software for heart rate variability analysis — https://www.kubios.com
- See also: information regarding heartmath sensor and application for heart rate variability data capture and analysis — https://www.heartmath.com